CLINICAL TRIAL: NCT02128256
Title: CERAMENT™|G - Bone Healing and Re-infection Prophylaxis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Olivier Borens (Other)
Responsible Party: Sponsor-Investigator, Dr. Olivier Borens, Head of Service of Traumatology and Septic Surgical Unit, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CeramentG-CH-2014
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; Bone substitute; Ceramic; Gentamicin
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cerament G injection (Experimental): Cerament G is injected to fill a bone defect after debridement of the infected bone.
  Interventions: Device: Cerament G

INTERVENTIONS:
Device: Cerament G

SUMMARY:
The surgical management of long bone infections is often challenging. Adequate surgical debridement decreases the bacterial load, removes dead tissues, and gives a chance for the host immune system and antibiotics to arrest infection. Adequate debridement may leave a large bony defect. An appropriate management of the dead space is essential to arrest the disease, and for maintenance of the bone's integrity. The current strategy includes the use of antibiotic-loaded bone cement that can be used to sterilize and temporarily maintain the dead space. The cement are usually removed after 2 to 4 weeks and replaced with a cancellous graft harvested from the hip of the patient.

CERAMENT™| G is a CE-marked resorbable ceramic bone graft substitute composed by calcium sulfate and calcium hydroxyapatite, intended to fill gaps and voids in the skeleton system and to promote bone healing. The antibiotic gentamicin is included in the ceramic to prevent colonization of gentamicin-sensible microorganisms in order to protect bone healing.

The aim of this study is to investigate the device absorption and bone in-growth of CERAMENT™| G in a surgically revised bone infection. In addition, bone healing and infection non-recurrence will be evaluated during 12 months of follow-up. The investigators expect a treatment success of >90 % and that a similar bone healing will be obtained as with a standard two-stage surgical procedure. In addition, the investigators believe that the use of CERAMENT™| G will be of advantage for the patient as bone healing will be achieved with a one-stage surgical procedure (in combination with antibiotic therapy), instead of a two-stage procedure, thus decreasing potential surgery-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a long bone infection in femur, tibia, humerus or radius
* Candidate for one stage procedure
* Patients above the age of 18
* Written informed consent obtained before any study-related activities
* Patients with communicative ability to understand the procedure and participate in the study and comply with the follow up program

Exclusion Criteria:

* Clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation
* Hypersensitivity to aminoglycoside antibiotics
* Myasthenia gravis
* Severe renal impairment
* Pre existing calcium metabolism disorder.
* Women who are pregnant or breastfeeding (a pregnancy test will be done in women of childbearing potential)
* History of hypersensitivity to the investigational device or any of its ingredients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Degree of device absorption after insertion of the device (during follow-up). | 3 and 12 months after surgery.
  The degree of device absorption will be evaluated by localized CT-scans 3 and 12 months after surgery.
Advances in bone in-growth after insertion of the device (during follow up). | 3 and 12 months after surgery.
  Bone in-growth will be evaluated by localized CT-scans 3 and 12 months after surgery.

SECONDARY OUTCOMES:
Bone healing | 6 weeks, 3 months, 6 months and 12 months after surgery.
  Bone healing will be evaluated by X-ray 6 weeks, 3 months, 6 months and 12 months after surgery.
Infection non-recurrence | During hospitalisation and 6 weeks, 3 months, 6 months and 12 months after surgery.
  Infection non-recurrence will be verified by measuring inflammatory blood parameters and body temperature, and through clinical examination (looking for pain, swelling, warmth and redness) during hospitalization (an expected average of 14 days following the surgery), and 6 weeks, 3 months, 6 months and 12 months after surgery (i.e. at each follow-up visit according to standard clinical praxis).
Serum gentamicin levels | 24 h, 48 h and 72 h after surgery.
  For evaluation of the gentamicin elution from the ceramic, serum gentamicin levels will be measured 24 h, 48 h and 72 h after surgery (during hospitalisation).

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Service of Orthopedy and Traumatology, Lausanne, Canton of Vaud, Switzerland